CLINICAL TRIAL: NCT01402011
Title: Rotator Cuff Tendinopathy: A Randomized and Blinded Comparison of Superficial and Deep Injection Methods
Brief Title: Study of 25% Dextrose Injections in Shoulder Ligaments and Tendons to Promote Their Healing
Acronym: Prolotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: WorkSafe BC (Unknown)
Responsible Party: Principal Investigator, Helene Bertrand, M.D., C.M, CCFP, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H09-00911; RS2010-OG07 (Other Grant/Funding Number: Worksafe BC)
Record Dates: First submitted 2011-06-20; First posted 2011-07-26 (Estimated); Results first posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Rotator Cuff Tendinitis
Keywords: Prolotherapy; regenerative injection therapy; dextrose injections
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Glucose; Prolotherapy; Lidocaine

STUDY DESIGN:
Intervention Model Description: Participants were randomly allocated into 3 groups to receive injections of 25% dextrose in .1% lidocaine or .1% lidocaine in the shoulder entheses, the 3rd group received .1% lidocaine subcutaneously above the shoulder entheses.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: For the 25% dextrose and .1% lidocaine and the .1% lidocaine enthesis injections, only the pharmacist knew the contents of each participant's numbered bottle. For the .1% subcutaneous injections, both the pharmacist and the physician where aware of the contents. There was a small c on the label. Only one participant asked the meaning of this letter, and he was told it stood for "contents".
Oversight: Data Monitoring Committee: No

ARMS (3):
- 25% dextrose in shoulder entheses (Experimental): 25% dextrose and .1% lidocaine injected in the shoulder entheses (ligament and tendon insertions on the periosteum).
  Interventions: Procedure: 25% dextrose in shoulder entheses
- .1% lidocaine in shoulder entheses (Active Comparator): .1% lidocaine injected in the shoulder entheses (ligament and tendon insertions on the periosteum).
  Interventions: Procedure: .1% lidocaine in shoulder entheses
- .1% lidocaine subcu. above shouldr enth. (Placebo Comparator): .1% lidocaine injected subcutaneously above the shoulder entheses (ligament and tendon insertions on the periosteum).
  Interventions: Procedure: .1% lidocaine subcu. above shouldr enth.

INTERVENTIONS:
Procedure: 25% dextrose in shoulder entheses — injections of 1 mL of 25% dextrose and .1% lidocaine solution in the following tendons: supraspinatus, infraspinatus, teres minor ( on greater tuberosity), subscapularis ( on lesser tuberosity), long tendon of biceps ( on supra-glenoid tubercle), short tendons of biceps on coracoid process, and the inferior glenohumeral ligament, anteriorly and posteriorly. If symptomatic the insertion of the teres minor and the triceps on the scapula.
  Other Names: Prolotherapy; regenerative injection therapy
  Arms: 25% dextrose in shoulder entheses
Procedure: .1% lidocaine in shoulder entheses — injections of 1 mL of .1% lidocaine 'ssolution in the following tendons: supraspinatus, infraspinatus, teres minor ( on greater tuberosity), subscapularis ( on lesser tuberosity), long tendon of biceps ( on supra-glenoid tubercle), short tendons of biceps on coracoid process, and the inferior glenohumeral ligament, anteriorly and posteriorly. If symptomatic the insertion of the teres minor and the triceps on the scapula.
  Other Names: Active control injections
  Arms: .1% lidocaine in shoulder entheses
Procedure: .1% lidocaine subcu. above shouldr enth. — injections of 1 mL of .1% lidocaine solution subcutaneously, above the following tendons: supraspinatus, infraspinatus, teres minor ( on greater tuberosity), subscapularis ( on lesser tuberosity), long tendon of biceps ( on supra-glenoid tubercle), short tendons of biceps on coracoid process, and the inferior glenohumeral ligament, anteriorly and posteriorly. If symptomatic, above the insertion of the teres minor and the triceps on the scapula.
  Other Names: Placebo injections
  Arms: .1% lidocaine subcu. above shouldr enth.

SUMMARY:
HYPOTHESIS: Prolotherapy, the injection of a growth promoting solution in injured ligaments and tendons of the shoulder is an effective treatment that decreases pain, increases functional capacity and promotes healing better and in less time than standard treatment with physiotherapy.

OVERVIEW: 75 subjects with rotator cuff tendinopathy proven by ultrasound will be recruited and assigned randomly into one of three groups of 25 to receive one of these three different treatments:

Group A (test): 25% dextrose with 0.1% lidocaine, injected into the tendons and ligaments Group B (control): 0.1% lidocaine injected in the rotator cuff tendons and ligaments Group C(control): 0.1% lidocaine injected subcutaneously above these structures All subjects will receive physiotherapy every other week for three months. To avoid placebo effects, patients, the radiologist and physiotherapist will not know to which treatment group the patients belong; the physician administering the injections will not be involved in assessing disability before or after treatment. (Note: The physician will know which patients belong to group C because it will be obvious: they are delivering a subcutaneous - versus a joint - injection).

There will be three sets of injections - one set per month for 3 months. The patients' condition will be tracked for nine months after the first treatment, to monitor changes in 3 outcome measures: pain (VAS and Rx #s), function (DASH and PESS), and tendon healing (as assessed by ultrasound).

DETAILED DESCRIPTION:
SAMPLE SIZE: Sample size justification: Dr. Bertrand reviewed 144 cases treated with prolotherapy, 25 of whom fit the inclusion criteria (between the ages of 19 and 74 and not suffering from arthritis of the shoulder or from frozen shoulder). Among those patients, the difference between the pain score prior to treatment and that when they were given the questionnaire averaged 5.36 points over10 with a standard deviation of 3.28. Improvements from baseline to 6 months on the true placebo arm were projected to be about half those of the prolotherapy group, averaging 2.7 points of improvement with a standard deviation approximately equal to that of the prolotherapy group of 3.28. In order to achieve an 80% power of detecting the differences in mean improvements, given each group has a standard deviation of 3.3, and the average difference between groups is 2.7 points out of 10, each group should include 25 subjects.

RECRUITMENT AND CONSENT:

Recruitment: Ads were sent to all the North Shore and Burnaby physicians, physiotherapists, and chiropractors, posted in the Lions gate hospital ultrasound waiting room and North Shore recreation centers. A small adwords ad referred subjects to our website, www.prolotherapyhealing/shoulder.

Consent: At the initial appointment with Dr. Bertrand, the patient will be given information about the nature of this study and the procedures involved, including the fact that each of three treatments will consist of numerous shoulder injections. He will also be told that up to three monthly treatments may be needed to achieve relief from shoulder pain. If he decides to proceed, he will be given a copy of the consent form, the DASH questionnaire, and the VAS pain scale to fill out. The intake assessment includes socio-demographic information and medical history including the duration and severity of symptoms, smoking status, arm dominance and general health. If the patient manifests symptoms and signs of a rotator cuff tendinopathy which has lasted more than three months, and has no exclusion criteria, he will be scheduled for an ultrasound and an x-ray examination of the shoulder. The radiologist will rate the ultrasound using the USPRS. If no exclusion criteria are found, the patient will be referred to the physiotherapist for a baseline assessment of his shoulder using the (PESS), and scheduled for his first treatment session. The patient will be told to avoid all anti-inflammatory medications for the four weeks following each treatment. He will be given a prescription of Tylenol three or Tramacet as needed for pain control.

RANDOM ALLOCATION OF PATIENTS, AND STUDY GROUPS:

At the first treatment session the patient will be assigned his sequential number. A previously generated master list will have randomly allocated each number either to treatment (A) or to one of two control groups (B), (C) using a permuted block randomization scheme. (The pharmacist will generate and have custody of the master list, using dice to ensure a random allocation.) Dr. Bertrand's file will record the patient's number. The pharmacist will prepare all the mixtures in advance and label them with the patient's number including the letter C, if the patient is to receive lidocaine subcutaneously.

Group A - intervention (treatment) group. Will receive three, monthly, prolotherapy session using a mixture of 25% dextrose and 0.1% lidocaine (50% dextrose mixed with equal parts of 0.2% lidocaine solution (one part 1% lidocaine mixed with four parts normal saline)) in the rotator cuff ligaments and tendons .

Group B - modified prolotherapy control group. Will receive a mixture 0.1% lidocaine (one part 1% lidocaine mixed with nine parts normal saline solution) in the rotator cuff ligaments and tendons.

Group C - true control group. Will receive 0.1% lidocaine (one part 1% lidocaine mixed with nine parts normal saline solution) subcutaneously above these same locations.

Intention to treat: Patients will be included in this study if they have received one set of injections. If, after the first treatment, they fail to keep their physician appointment, the secretary will telephone the patients and administer the DASH questionnaire and the VAS by phone. She will do this according to the study timeline (i.e. one, two, three and six months following their first injection session).

INTERVENTION PROTOCOL: Injection procedure. After patients are randomized to Groups A, B, and C, they will receive three sets of injections (one set per month for 3 months). The entire shoulder area will be sterilized with 70% alcohol. In order to decrease the pain of the actual injections, the areas to be treated will be injected intradermally, using a number 32G one half inch needle, with a mixture of 1% Xylocaine buffered by an equal volume of sodium bicarbonate solution for both subjects and controls. The intervention will consist of the following: For groups A and B, the solution will be injected, in 1 mL amounts, using a 27G 1½ to two inch needle in the following locations:

Supraspinatus tendon: on the anterior-superior part of the greater tuberosity, this tendon is generally tender to palpation over an area of about 2 to 3 cm in height and 1 cm in width. Unless the tendon is tender to palpation, 1 mL of solution is injected. All tender parts of the tendon are injected at 1 cm intervals, each with .5 mL of solution, a total of 1 to four injections.

Infraspinatus tendon: immediately posterior to the supraspinatus tendon, it is in line with the spine of the scapula on the greater tuberosity. Unless the tendon is tender to palpation, 1 mL of solution is injected. All tender parts of the tendon are injected at 1 cm intervals, each with .5 mL of solution, a total of 1 to four injections.

Teres minor tendon: attaches on the posterior superior surface of the greater tuberosity. Unless the tendon is tender to palpation, 1 mL of solution is injected. All tender parts of the tendon are injected at 1 cm intervals, each with .5 mL of solution, a total of 1 to four injections.

Teres minor and triceps insertion on the outer edge of the scapula. To avoid the risk of injecting the lungs, the injections are made with the subject's arm in extreme adduction, as if to scratch his back. This brings the scapula forward, distancing it from the rib cage. These areas are injected only if the subject complains of tenderness to palpation. All tender areas are injected at 1 cm intervals, each with .5 mL of solution, a total of 1 to four injections.

Coracoid process: insertion of the short tendon of the biceps. It is the bony pro-eminence under the clavicle medial to the head of the humerus. 1 mL of solution is injected in the area.

Long tendons of biceps: immediately medial to the acromioclavicular joint, with the arm in slight external rotation a 2 inch needle is inserted vertically with a 15° anterior tilt until bone is reached. 1 mL of solution is injected in the area.

Subscapularis tendon: inserts on the lesser tuberosity of the humerus posterior to the long tendon of the biceps. With the arm in full external rotation and adduction, a 2 inch needle is inserted 1 cm lateral to the coracoid process until it reaches the humerus. 1 mL of solution is injected in the area. Additional injections can be performed 1 cm above and 1 cm below this area with .5 mL of solution if the subscapularis is tender to palpation.

Inferior glenohumeral ligament: with the arm externally rotated and abducted 90°, a 2 inch needle is inserted posteriorly 1 cm below the coracoid process until the inferior part of the glenohumeral joint is reached. 1 mL is inserted in the area and the needle is moved medially and laterally. Another milliliter is injected in each of those two areas, corresponding to the scapular and humeral insertion of the inferior glenohumeral ligament. 22G, 3 or 4 inch needles are used for obese subjects.

All needle insertions are made until bone is reached. No injection is done otherwise.

At the end of the procedure, the entire shoulder joint should be pain free and exhibit full or almost full range of motion. The patient will be warned that this pain free status will only last as long as the local anesthetic is in place.

The control group (Group C) will be treated in all respects identically to groups A and B, with the following exceptions: (1) they will receive injections of 0.1% lidocaine combined with normal saline (unlike group A), and (2) the depth of the injections will be different, subcutaneous rather than inside the ligaments, but the same volume of solution will be used as for groups A and B.

To assess if the subjects are truly blind as to their treatment, they will be asked to state which treatment (true prolotherapy, modified prolotherapy, placebo, don't know) they think they have received after each treatment, and this will be recorded on the patient's chart and database. Neither the patient nor the physiotherapist or radiologist will be aware to which group the patient has been randomized.

Outcome measures assessment: At each of the 3 treatment sessions, we will: (1) record side effects experienced during the session or following the previous injection session, and (2) administer the VAS pain scale, and DASH (disabilities of the arm, shoulder and hand) questionnaire prior to being treated. If requested, patients will receive a prescription for either Tylenol number three or Tramacet to deal with post-treatment pain. The amounts prescribed and the amounts used will be recorded.

Throughout the 3-month injection intervention, subjects will also receive physiotherapy every 2 weeks. One month and 3 months after the third set of injections patients will be reassessed by the physiotherapist using the (PESS) and also fill out the VAS pain scale and answer the DASH questionnaire. Finally, a follow-up ultrasound (USPRS) will be administered 3 months after completing the injections.

Nine months after treatment started: follow-up telephone survey, to determine whether improvements are retained.

STATISTICAL ANALYSIS:

With the exception of 'total amount of pain medication used', the main assessment for each of the outcome measures (VAS, DASH, PESS, USPRS), will be based on the difference in each patient's scores from their first (baseline) visit to their last visit six months later. For each outcome, the three groups will be compared using ANOVA. In cases where the ANOVA indicates differences between the three groups, subsequent comparisons of the prolotherapy group to each of the control groups will be carried out. The overall primary assessment is the comparison of the prolotherapy group (A) to the true control group (C) on the VAS improvements from baseline to six months; all other analyses are secondary. All statistical tests will be two-sided and differences will be considered statistically significant if the p-value is less than 0.05.

To further explore the pattern of the treatment effect over time, the improvements from baseline to other time points will be analyzed similarly. Methods of longitudinal data analysis will be used to carry out more comprehensive exploratory analyses.

Other variables, collected at the first patient visit, such as duration of pain prior to randomization, the patient's age and gender, their general health and smoking status, whether the tendinopathy affects the dominant arm, and the severity of the tendinopathy can influence the duration and intensity of pain, shoulder function, and ultrasound evidence of healing. The relationships of such prognostic factors with the outcome measures will be examined. In cases where strong relationships are apparent, the above analyses will be repeated with adjustment for such factors. That is, the analysis of covariance (ANCOVA) will be used in place of ANOVA, with the corresponding subsequent comparisons of the prolotherapy group to each of the control groups.

SIGNIFICANCE:

Rotator cuff tendinopathy is known to be notoriously resistant to standard therapy using NSAIDs, physiotherapy, steroid injections and surgery. After three years only 46% are pain-free. In my experience, using prolotherapy, 75% are more than 50% improved after three months, at which time 42% are pain-free. If this experience is corroborated by the current research project, this may augur a radical change in the way rotator cuff tendinopathy is treated. The materials needed for prolotherapy ( syringes, needles, dextrose solution and local anesthetic) are inexpensive and available to all family practitioners regardless of their location. The knowledge needed is relatively easy for family physicians to acquire, making this treatment potentially accessible even in the remotest rural locations where surgery and even physiotherapy are unavailable. There are no major nerves or blood vessels in the areas injected, so the risks of this treatment are extremely low (e.g. bruising and soreness for a few days following the injections. These complications compare favorably with the 10% complication rate following shoulder surgery, which also requires a prolonged postoperative recovery period, and the, at times serious, potential side effects of NSAIDs and corticosteroid injections. Getting people to return to work sooner, and for much less cost than the current therapies (3x $150 compared to $24,300) would benefit both the healthcare system and those who suffer with this problem.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients over 19 and less than 75 years of age

Exclusion Criteria:

* allergy to corn, as the dextrose solution is corn-based
* allergy to local anesthetic
* immune deficiency
* conditions requiring anti-inflammatory medications including prednisone, corticosteroid injection less than eight weeks prior to the first set of injections
* use of immune suppressants
* symptomatic osteoarthritis of the gleno-humeral or acromio-clavicular joint
* age over 75 or under 19
* adhesive capsulitis based on a thorough physical examination, where shoulder flexion or abduction is below 100 °, horizontal adduction is below 30 °, the hand behind the back is below the waist, external rotation is less than 30 °
* full thickness tear greater than 1.2 cm as seen on ultrasound
* autoimmune disorders such as lupus or rheumatoid arthritis
* neurological disorders including Parkinson, seizures, and dementias are excluded for patient safety during the procedures
* HIV, viral hepatitis and other blood borne communicable diseases, to protect the investigators
* calcium deposits greater than 8 mm in diameter
* type III acromion as seen on x-ray
* painful condition elsewhere in the body likely to cloud the subject's assessment of his shoulder pain
* no evidence of tendinopathy as seen on ultrasound
* uncontrolled diabetes: A1C > 7

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helene Bertrand, MD, CCFP, Principal Investigator — University of British Columbia, Vancouver Coastal Health Research Institute
Locations (2):
- Canada (2):
  - Dr. Helene Bertrand Inc., 220-1940 Lonsdale Avenue, North Vancouver, British Columbia
  - Active shoulder clinics, West Vancouver sports and orthopedic physiotherapy, 210- 575 16th Street, West Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Yes
The de-identified database Is now available on request to Doctor Helene Bertrand at heleneb@mail.UBC.ca
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available from January 2015 to January 2020
Access Criteria: This study was published in Archives Of Physical Medicine And Rehabilitation 2016 volume 97 pages 17 - 25 under the title: Dextrose Prolotherapy Versus Control Injections In Painful Rotator Cuff Tendinopathy

REFERENCES:
- [Background] Coombes BK, Bisset L, Vicenzino B. Efficacy and safety of corticosteroid injections and other injections for management of tendinopathy: a systematic review of randomised controlled trials. Lancet. 2010 Nov 20;376(9754):1751-67. doi: 10.1016/S0140-6736(10)61160-9. Epub 2010 Oct 21. PMID 20970844
- [Background] Silverstein B, Welp E, Nelson N, Kalat J. Claims incidence of work-related disorders of the upper extremities: Washington state, 1987 through 1995. Am J Public Health. 1998 Dec;88(12):1827-33. doi: 10.2105/ajph.88.12.1827. PMID 9842381
- [Background] Stovitz SD, Johnson RJ. NSAIDs and musculoskeletal treatment: what is the clinical evidence? Phys Sportsmed. 2003 Jan;31(1):35-52. doi: 10.3810/psm.2003.01.160. PMID 20086440
- [Background] Cohen DB, Kawamura S, Ehteshami JR, Rodeo SA. Indomethacin and celecoxib impair rotator cuff tendon-to-bone healing. Am J Sports Med. 2006 Mar;34(3):362-9. doi: 10.1177/0363546505280428. Epub 2005 Oct 6. PMID 16210573
- [Background] Gaujoux-Viala C, Dougados M, Gossec L. Efficacy and safety of steroid injections for shoulder and elbow tendonitis: a meta-analysis of randomised controlled trials. Ann Rheum Dis. 2009 Dec;68(12):1843-9. doi: 10.1136/ard.2008.099572. Epub 2008 Dec 3. PMID 19054817
- [Background] Lewis JS. Rotator cuff tendinopathy/subacromial impingement syndrome: is it time for a new method of assessment? Br J Sports Med. 2009 Apr;43(4):259-64. doi: 10.1136/bjsm.2008.052183. Epub 2008 Oct 6. PMID 18838403
- [Background] Mansat P, Cofield RH, Kersten TE, Rowland CM. Complications of rotator cuff repair. Orthop Clin North Am. 1997 Apr;28(2):205-13. doi: 10.1016/s0030-5898(05)70280-7. PMID 9113716
- [Background] Brislin KJ, Field LD, Savoie FH 3rd. Complications after arthroscopic rotator cuff repair. Arthroscopy. 2007 Feb;23(2):124-8. doi: 10.1016/j.arthro.2006.09.001. PMID 17276218
- [Background] Liu X, Luo F, Pan K, Wu W, Chen H. High glucose upregulates connective tissue growth factor expression in human vascular smooth muscle cells. BMC Cell Biol. 2007 Jan 16;8:1. doi: 10.1186/1471-2121-8-1. PMID 17224075
- [Background] Fullerton BD. High-resolution ultrasound and magnetic resonance imaging to document tissue repair after prolotherapy: a report of 3 cases. Arch Phys Med Rehabil. 2008 Feb;89(2):377-85. doi: 10.1016/j.apmr.2007.09.017. PMID 18226666
- [Background] K. Dean Reeves, MD; Bradley D. Fullerton, MD, FAAPMR and Gaston Topol, MD Evidence-Based Regenerative Injection Therapy (Prolotherapy)in Sports Medicine sports Medicine Resource Manual 2008 Chapter 50.
- [Background] Scarpone M, Rabago DP, Zgierska A, Arbogast G, Snell E. The efficacy of prolotherapy for lateral epicondylosis: a pilot study. Clin J Sport Med. 2008 May;18(3):248-54. doi: 10.1097/JSM.0b013e318170fc87. PMID 18469566
- [Background] Reeves KD, Hassanein K. Randomized prospective double-blind placebo-controlled study of dextrose prolotherapy for knee osteoarthritis with or without ACL laxity. Altern Ther Health Med. 2000 Mar;6(2):68-74, 77-80. PMID 10710805
- [Background] Reeves KD, Hassanein K. Randomized, prospective, placebo-controlled double-blind study of dextrose prolotherapy for osteoarthritic thumb and finger (DIP, PIP, and trapeziometacarpal) joints: evidence of clinical efficacy. J Altern Complement Med. 2000 Aug;6(4):311-20. doi: 10.1089/10755530050120673. PMID 10976977
- [Background] David Rabago Prolotherapy for chronic musculoskeletal pain Complementary and alternative therapies in the aging population edited by Ronald Ross Watson chapter 2 15-44 Elsevier 2009
- [Result] Bertrand H, Reeves KD, Bennett CJ, Bicknell S, Cheng AL. Dextrose Prolotherapy Versus Control Injections in Painful Rotator Cuff Tendinopathy. Arch Phys Med Rehabil. 2016 Jan;97(1):17-25. doi: 10.1016/j.apmr.2015.08.412. Epub 2015 Aug 22. PMID 26301385

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2010 and April 2012 advertisements for those between 19 and 75 years, with shoulder pain greater than 3 months, were placed in tennis courts, gymnasia, the Lions Gate Hospital Ultrasound Department, and sent to local physicians.
Pre-assignment Details: Clinical check R/O:unqualified participants. 77 were probable participants, pending results from their diagnostic ultrasound (delayed treatment period). 77 were ultimately enrolled in the study.
Groups:
- 25% Dextrose in Ligaments and Tendons: 25% dextrose and .1% lidocaine injected in the rotator cuff ligaments and tendons.
  shoulder injections: injections of 1 mL of solution in the following tendons: supraspinatus, infraspinatus, teres minor ( on greater tuberosity), subscapularis ( on lesser tuberosity), long tendon of biceps ( on supra-glenoid tubercle), short tendons of biceps on coracoid process, and the inferior glenohumeral ligament, anteriorly and posteriorly. If symptomatic the insertion of the teres minor and the triceps on the scapula.
- .1% Lidocaine in Ligaments and Tendons: .1% lidocaine injected in the shoulder ligaments and tendons
  shoulder injections: injections of 1 mL of solution in the following tendons: supraspinatus, infraspinatus, teres minor ( on greater tuberosity), subscapularis ( on lesser tuberosity), long tendon of biceps ( on supra-glenoid tubercle), short tendons of biceps on coracoid process, and the inferior glenohumeral ligament, anteriorly and posteriorly. If symptomatic the insertion of the teres minor and the triceps on the scapula.
- .1% Lidocaine Subcutaneous: .1% lidocaine injected subcutaneously above the ligaments and tendons of the shoulder.
  shoulder injections: injections of 1 mL of solution subcutaneously above the following tendons: supraspinatus, infraspinatus, teres minor ( on greater tuberosity), subscapularis ( on lesser tuberosity), long tendon of biceps ( on supra-glenoid tubercle), short tendons of biceps on coracoid process, and the inferior glenohumeral ligament, anteriorly and posteriorly. If symptomatic above the insertion of the teres minor and the triceps on the scapula.
Period: Delayed Treatment Period
Arm/Group | 25% Dextrose in Ligaments and Tendons | .1% Lidocaine in Ligaments and Tendons | .1% Lidocaine Subcutaneous
Started | 29 | 23 | 26
Completed | 28 (One patient with needle phobia declined to be treated before the 1st set of injections) | 23 | 26
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Active Treatment Period
Arm/Group | 25% Dextrose in Ligaments and Tendons | .1% Lidocaine in Ligaments and Tendons | .1% Lidocaine Subcutaneous
Started | 28 | 23 | 26
Completed (Patients who quit the study did so because they found the injections too painful.) | 27 | 20 | 26
Not Completed | 1 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0
Period: Nine Month Follow-up
Arm/Group | 25% Dextrose in Ligaments and Tendons | .1% Lidocaine in Ligaments and Tendons | .1% Lidocaine Subcutaneous
Started | 27 | 20 | 26
Completed | 27 | 19 | 26
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 25% Dextrose in Ligaments and Tendons | .1% Lidocaine in Ligaments and Tendons | .1% Lidocaine Subcutaneous | Total
Number analyzed (Participants) | 27 | 20 | 26 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (13.5) | 51.1 (9.2) | 49.0 (11.9) | 51 (11.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 10 | 27
  Male | 16 | 14 | 16 | 46
Shoulder symptom duration [Mean (Standard Deviation); unit: months] | 61 (81) | 131 (155) | 101 (115) | 76 (166)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Pain Scale 0= no Pain 10 = Maximum Pain
Description: Subject marks his pain level at rest, at work, doing sports on a 10 cm scale. The maximum pain level among the 3 different activities was recorded.
Time Frame: 20 minutes before first injection on first day of patient visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 25% Dextrose in Shoulder Entheses | .1% Lidocaine in Shoulder Entheses | .1% Lidocaine Subcu. Above Shouldr Enth.
Number analyzed (Participants) | 27 | 19 | 26
units on a scale | 7.3 (0.4) | 6.9 (0.5) | 6.9 (0.4)

2. Primary Outcome: Change From Baseline of Visual Analog Pain Scale at 3 Months
Description: Subject marks his pain level at rest, at work, doing sports on a 10 cm scale. Maximum of pain scores rest, work, sport recorded. Calculated as pain at baseline - pain at 3 months. VAS scale is from 0 = no pain to 10 = maximum pain
Time Frame: baseline and three months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 25% Dextrose in Ligaments and Tendons | .1% Lidocaine in Ligaments and Tendons | .1% Lidocaine Subcutaneous
Number analyzed (Participants) | 27 | 19 | 26
units on a scale | 3.0 (0.5) | 2.7 (0.7) | 2.7 (0.6)

3. Primary Outcome: Change From Baseline in Maximum Pain Score at 9 Months
Description: Participants were asked about pain at rest, at work, doing sports. The maximum pain reported on a scale ranging from 0 (no pain at all) to 10 (extreme pain) was recorded for each participant. Maximum of pain scores rest, work, sport recorded. Calculated as pain at baseline - pain at 9 months.
Time Frame: baseline and 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 25% Dextrose in Ligaments and Tendons | .1% Lidocaine in Ligaments and Tendons | .1% Lidocaine Subcutaneous
Number analyzed (Participants) | 27 | 19 | 26
units on a scale | 2.9 (0.6) | 1.8 (0.7) | 1.3 (0.6)

4. Secondary Outcome: Rotator Cuff Ultrasound, Ultrasound Shoulder Pathology Rating Scale
Description: From Brose et al. "shoulder ultrasound abnormalities, physical examination findings, and pain in manual wheelchair users with spinal cord injury" Arch Phys Med Rehabil 2008 Nov, 89: 2086-93 appendix 2. rates biceps tendinopathy (0-6), supraspinatus tendinopathy (0-5), greater tuberosity the cortical surface (0-3), dynamics supraspinatus impingement (0-3), dynamic subscapularis/ biceps/ coracoid impingement (0-3). The total score ranged from 0 to 20 with higher scores indicating a worse outcome. The change was calculated by taking the final score - the baseline score.
Time Frame: 20 minutes before first injection on first day of patient visit and at on average 9.4 months
Population: Three of the 25% dextrose in ligaments and tendons group did not show up for their ultrasound appointment at nine months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 25% Dextrose in Ligaments and Tendons | .1% Lidocaine in Ligaments and Tendons | .1% Lidocaine Subcutaneous
Number analyzed (Participants) | 24 | 19 | 26
units on a scale
  Baseline | 4.0 (0.4) | 4.3 (0.5) | 4.3 (0.4)
  change at 9.4 +/- 2.2 months | -0.3 (0.5) | -0.6 (0.5) | -0.6 (0.4)

5. Secondary Outcome: Physical Examination of the Shoulder Scale
Description: From Steven W. Brose, DO, Michael L. Boninger, MD, Bradley Fullerton, MD, Thane McCann, MD, From: Jennifer L. Collinger, BSE, Bradley G. Impink, BSE, Trevor A. Dyson-Hudson, MD Shoulder ultrasound abnormalities, physical examination findings, and pain in manual wheelchair users with spinal cord injury. Arch Phys Med Rehabil 2008 Nov; 89:2086-93, appendix 1 12 parameters of shoulder examination: Biceps tendon/bicipital groove tenderness, Supraspinatus tendon/greater tuberosity tenderness Acromioclavicular joint tenderness Resisted external rotation. Resisted internal rotation. Supraspinatus test. Painful Arc Test. Neer impingement sign. Hawkins-Kennedy impingement sign. O'Brien Active Compression Test for AC Joint Pathology O'Brien Active Compression Test for Labral Pathology impingement sign. each test scored 0 = no pain, 1 = tenderness, 2 = pain. All 12 scores added. Range 0-24. Higher scores = more pathology
Time Frame: 20 minutes before first injection on first day of patient visit and at 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 25% Dextrose in Ligaments and Tendons | .1% Lidocaine in Ligaments and Tendons | .1% Lidocaine Subcutaneous
Number analyzed (Participants) | 27 | 19 | 26
units on a scale
  Baseline | 13.2 (4.8) | 13.1 (3.7) | 13 (3.5)
  3 months | 11.4 (5.6) | 10.7 (5.3) | 12.9 (3.9)

6. Secondary Outcome: Disabilities of the Arm Shoulder and Hand Questionnaire
Description: http://www.dash.iwh.on.ca/assets/images/pdfs/DASH_quest06.pdf 30 questions assessing ability to use shoulder in everyday activities, each question scored 1 to 5, where one is normal, no problem and five is unable to perform. No data was collected at 9 months. The score ranges from 30 to 150. Higher scores represent worse outcomes.
Time Frame: 20 minutes before the first injection and at 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 25% Dextrose in Ligaments and Tendons | .1% Lidocaine in Ligaments and Tendons | .1% Lidocaine Subcutaneous
Number analyzed (Participants) | 27 | 19 | 26
units on a scale
  Baseline | 72.4 (21.6) | 71.3 (19.4) | 69.6 (22.9)
  3 months | 61.3 (17.2) | 54.7 (16.2) | 61 (18.4)

7. Secondary Outcome: Nine Month Satisfaction Questionnaire
Description: Phone call asking how satisfied were they with their treatment 10 = extremely satisfied, 0 = extremely dissatisfied )
Time Frame: Nine months after first injection treatment appointment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 25% Dextrose in Ligaments and Tendons | .1% Lidocaine in Ligaments and Tendons | .1% Lidocaine Subcutaneous
Number analyzed (Participants) | 27 | 19 | 26
units on a scale | 6.7 (3.2) | 4.7 (4.1) | 3.9 (3.1)

8. Other Pre Specified Outcome: Total Prescription Pain Medication Used
Description: Total amount of narcotic pain medication prescribed. Data were not collected at 1,2,3 and 6 months.
Time Frame: 20 minutes before first injection on first day of patient visit
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Visual Analog Pain Scale
Description: Subject marks his pain level at rest, at work, doing sports on a 10 cm scale.
Time Frame: two months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Visual Analog Pain Scale
Description: Subject marks his pain level at rest, at work, doing sports on a 10 cm scale. Maximum of pain scores rest, work, sport is recorded.
Time Frame: one month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- .1% Lidocaine Subcutaneous: .1% lidocaine injected subcutaneously above the ligaments and tendons of the shoulder.
  shoulder injections: injections of 1 mL of solution in the following tendons: supraspinatus, infraspinatus, teres minor ( on greater tuberosity), subscapularis ( on lesser tuberosity), long tendon of biceps ( on supra-glenoid tubercle), short tendons of biceps on coracoid process, and the inferior glenohumeral ligament, anteriorly and posteriorly. If symptomatic the insertion of the teres minor and the triceps on the scapula.
Arm/Group | 25% Dextrose in Ligaments and Tendons | .1% Lidocaine in Ligaments and Tendons | .1% Lidocaine Subcutaneous
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/20 | 0/26
Other Adverse Events (participants affected / at risk) | 0/27 | 1/20 | 0/26
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25% Dextrose in Ligaments and Tendons (N=27) | .1% Lidocaine in Ligaments and Tendons (N=20) | .1% Lidocaine Subcutaneous (N=26)
Frozen Shoulder Development (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — One participant developed frozen shoulder injection after injection. This participant was referred for additional physical therapy with resolution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No